CLINICAL TRIAL: NCT02477865
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase IIIa Clinical Study Evaluating PEGylated Loxenatide Injection（PEX168）in Monotherapy of Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of PEX168 in Monotherapy Diabetes Mellitus Type 2 Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEX168-301
Record Dates: First submitted 2015-05-28; First posted 2015-06-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — polyethylene glycol loxenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEX168(100µg) (Experimental): PEX168(100µg),100µg,Subcutaneous injection,once a week,for 52 weeks.
  Interventions: Drug: PEX168(100µg)
- PEX168(200µg) (Experimental): PEX168(200µg),200µg,Subcutaneous injection,once a week,for 52 weeks.
  Interventions: Drug: PEX168(200µg)
- Placebo (Placebo Comparator): Placebo,0.5ml,Subcutaneous injection,once a week for 24 weeks,followed by PEX168(100µg or 200µg) qw sc for 28 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PEX168(100µg) — 100µg,Subcutaneous injection,once a week. continued for 52 weeks
  Other Names: Polyethylene Glycol Loxenatide
  Arms: PEX168(100µg)
Drug: PEX168(200µg) — 200µg,Subcutaneous injection,once a week. continued for 52 weeks
  Other Names: Polyethylene Glycol Loxenatide
  Arms: PEX168(200µg)
Drug: Placebo — 0.5ml,Subcutaneous injection,once a week.continued for 24 weeks,then use PEX168 100µg or 200µg qw sc.for 28 weeks.
  Other Names: Injection mimetic
  Arms: Placebo

SUMMARY:
This is a phase III, multicenter, randomized, double-blind, placebo-controlled study planning to include approximately 387 T2DM patients who have received at least 8 weeks of treatment with diet control and exercise； have not received any glucose-lowering agents within the 8 weeks prior to screening; and have inadequately controlled blood glucose.The subjects would receive PEX168 or placebo monotherapy for 52weeks in total.

DETAILED DESCRIPTION:
This study consists of 4 periods： Period 1：Up to 3 weeks of screening period. Period 2：A 4-week PEX168 dummy run-in period. Period 3：A 52-week treatment period (including a 24-week core treatment period and a 28-week extended treatment period).

Period 4: A 4-week safety follow-up period. This study will last for approximately 63 weeks, including up to approximately 60 clinic visits.

ELIGIBILITY:
Inclusion Criteria (all of the 8 must be met)：

1. Type 2 diabetes mellitus confirmed by the 1999 WHO criteria；
2. Men or women；
3. Age at signing the ICF≥18 years and ≤78 years；
4. Body mass index (BMI) 20-40 Kg/m2；
5. At least 8 weeks of treatment with diet control and exercise received prior to screening；
6. No glucose-lowering agents received within the 8 weeks prior to screening；
7. 7.5%≤HbA1c≤11.0% at screening（local or centralized test）； 7.0%≤HbA1c≤10.5% at randomization（centralized test），and FBG< 13.9 mmol/L（local test）；
8. Ability to understand the procedures and approach of this study, willingness to complete the study in strict compliance with the protocol and to voluntarily sign the ICF.

Exclusion criteria：

1. Investigator suspecting the subject of allergy to the study drug；
2. Use of any of the following medications or therapies prior to screening：

   1. GLP-1 receptor agonists, GLP-1 analogues, DPP-4 inhibitors or any other incretin analogues.
   2. Growth hormone therapy within the 6 months prior to screening；
   3. History of drug abuse or alcohol abuse；
   4. Participation in any clinical trial within the 3 months prior to screening；
   5. Prolonged intravenous, oral or intraarticular treatment with corticosteroids within the 2 months prior to screening;
   6. Use of any weight control agents or surgeries within the 2 months prior to screening;
   7. Any medications used prior to screening that at the investigator's discretion may confound the interpretation of the efficacy or safety data；
3. History or evidence of any of the following conditions prior to screening：

   1. Type 1 diabetes mellitus, single gene mutation DM, DM associated with pancreatic injury，or secondary DM；
   2. History of hypertension with SBP>160 mmHg and/or DBP>100 mmHg；
   3. History of acute/chronic pancreatitis, history of symptomatic cholecystopathy;
   4. History of myeloid C-cell carcinoma, history of multiple endocrine neoplasm （MEN） 2A or 2B syndrome, or related familiar history；
   5. Gastric emptying disorders, severe chronic gastrointestinal disorders;
   6. History of severe hypoglycemia, unconsciousness or severe hypoglycemia history；
   7. Significant hematological disorders, or any diseases；
   8. Severe diabetic complications that in the opinion of the investigator make the subject not suitable to participate in this study；
   9. Tumors of any organ or system that not been treated within the 5 years prior to screening；
   10. Coronary angioplasty, coronary stenting, coronary artery bypass, uncompensated heart failure （NYHA Class III or IV）, within the 6 months prior to screening；
   11. Acute metabolic complications within the 6 months prior to screening；
   12. Thyroid dysfunction within the 6 months prior to screening；
   13. Blood lipid disorders within the 6 months prior to screening；
   14. Any severe trauma or severe infection within the 1 month prior to screening；
4. Laboratory indicators meeting any of the following criteria prior to screening：

   1. ALT>2.5×ULN and/or AST>2.5×ULN and/or total bilirubin>2.5×ULN；
   2. Hemoglobin≤100 g/L；
   3. Serum creatinine>1.5×UNL and eGFR < 45 ml/min/1.73 m2； eGFR is calculated as：186.3 ×[（Serum Creatinine（mmol/L）/88.4）]-1.154 × [Age (years)]- 0.203 × 1.223 × 0.742 （Females） or ×1（Males）
   4. Serum thyroid-stimulating hormone（TSH） out of the reference range that is assessed as clinically significant by the investigator;
   5. Fasting TGL>5.64 mmol/L（500 mg/dl）；
   6. Blood amylase and urine amylase>ULN that is assessed as clinically significant by the investigator；
   7. Any clinically significant laboratory abnormalities；
5. Clinically significant 12-lead ECG abnormalities；
6. Blood donation or loss≥400 mL，or receipt of blood donation within the 4 weeks prior to screening；
7. Pregnant or lactating women, or men or women of child-bearing potential not willing to take contraceptive measures during the study；
8. Any other conditions of the subject that at the investigator's discretion may compound the interpretation of the efficacy or safety data.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2014-03-23 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseling to 24 weeks
  To evaluate the HbA1c change from baseline to treatment Week 24 when receiving PEX 168 as compared to the placebo, given on the basis of diet control and exercise.

SECONDARY OUTCOMES:
The proportion of HbA1c <6.5% and <7% at the end of the analysis. | Baseling to 24 weeks
  The proportion of HbA1c <6.5% and <7% at the end of the analysis, and the proportion receiving salvage therapy.
Fasting plasma glucose | Baseling to 52 weeks
6 points glucose of fingertip | Baseling to 24 and 52 weeks
  Each test point of time was before breakfast, 2 hours after breakfast, before lunch,2 hours after lunch , dinner, 2 hours after dinner.This test was performed four times including baseline,V19,V31 and V59.
Postprandial blood glucose two hours | Baseling to 24 weeks
Postprandial blood glucose two hours AUC | Baseling to 24 weeks
Lipid | Baseling to 52 weeks
Weight measured by standardized procedure. | Baseling to 52 weeks
  Collect weight data in the morning of screening period, baseline,4,8,12,18,24,38,52 weeks by standardized procedure.
Blood pressure | Baseling to 52 weeks
  Collect blood pressure data in the morning of screening period, baseline,4,8,12,18,24,38,52 weeks by standardized procedure.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseling to 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenying Yang, MD, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No